CLINICAL TRIAL: NCT02557477
Title: Omega 3/6 Fatty Acids for Reading in Children: A Randomised, Double-blind, Placebo-controlled Trial in 9-year-old Mainstream Schoolchildren in Sweden
Brief Title: Omega 3/6 Fatty Acids for Reading in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 381-09
Record Dates: First submitted 2015-09-13; First posted 2015-09-23 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Reading Ability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Participants received 3 capsules of Omega 3/6 fatty acids twice daily
  Interventions: Dietary Supplement: Omega 3/6 fatty acids
- Placebo (Placebo Comparator): Participants received 3 capsules of identical placebo (palm oil) twice daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega 3/6 fatty acids — Three Omega 3/6 capsules twice daily
  Arms: Active
Dietary Supplement: Placebo — Three placebo capsules twice daily
  Arms: Placebo

SUMMARY:
The primary objective was to assess whether supplementation of Omega 3/6 fatty acids improves mainstream schoolchildren's reading ability. The secondary objective was to assess whether Omega 3/6 improves cognitive functions such as attention, memory, learning, language/communication, problem solving and social ability.This was a 3-month randomised, double-blind, placebo-controlled study followed by one-way crossover (placebo to active treatment) for an additional 3 months. Mainstream schoolchildren aged 9-10 years were initially randomised to receive three Omega 3/6 capsules twice daily or identical placebo. All outcome measures were assessed at baseline, 3 months and 6 months. The primary outcome measure was the LOGOS test, a comprehensive test battery for evaluating reading abilities. Secondary outcome measures were the parent-rated Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale-IV, 5-15 scale (domains of learning, memory, language/communication and problem solving); Social and Communication Disorders Checklist (to evaluate social ability)

DETAILED DESCRIPTION:
This was a 3-month randomized, double-blind, placebo-controlled study (Period 1) followed by one-way crossover (placebo to active treatment) for an additional 3 months (Period 2). Participants were randomized to receive three Omega 3/6 capsules twice daily (corresponding to a daily dose of 558 mg EPA, 174 mg DHA, and 60 mg gamma-linolenic acid) or identical placebo capsules (palm oil). All daily doses were taken at home supervised by the parents. All outcome measures were assessed at baseline and at the 3- and 6-month follow-up visits. The participants were mainstream schoolchildren in the 3rd school year (aged 9-10 years). Exclusion criteria were continuous supplementation of Omega-3 fatty acids for periods longer than 1 month during the previous year, significant medical conditions (e.g. diabetes, epilepsy), intellectual disability, attention-deficit hyperactivity disorder (ADHD) diagnosis, psychoactive medication, or substance use.

ELIGIBILITY:
Inclusion Criteria:

* mainstream schoolchildren in the 3rd school year (aged 9-10 years).

Exclusion Criteria:

* continuous supplementation of Omega-3 fatty acids for periods longer than 1 month during the previous year
* significant medical conditions (e.g. diabetes, epilepsy)
* intellectual disability
* attention-deficit hyperactivity disorder (ADHD) diagnosis, psychoactive medication, or substance use.

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in reading ability | 0, 3 and 6 months
  LOGOS test: Computerized test of several functions implicated in reading ability

SECONDARY OUTCOMES:
Change in ADHD symptom severity | 0, 3 and 6 months
  ADHD-Rating Scale IV: Parent-rated questionnaire measuring the DSM-IV ADHD symptom criteria
Change in learning ability | 0,3 and 6 months
  FTF scale: Parent-rated questionnaire, domain measuring problem scores in learning ability
Change in memory ability | 0, 3 and 6 months
  FTF scale: Parent-rated questionnaire, domain measuring problem scores in memory ability
Change in language/communication ability | 0,3 and 6 months
  FTF scale: Parent-rated questionnaire, domain measuring problem scores in language/communication ability
Change in problem solving ability | 0,3 and 6 months
  FTF scale: Parent-rated questionnaire, domain measuring problem scores in problem solving ability
Change in social ability | 0,3 and 6 months
  Social and Communication Disorders Checklist (SCDC): Parent-rated checklist measuring social ability

REFERENCES:
- [Derived] Johnson M, Fransson G, Ostlund S, Areskoug B, Gillberg C. Omega 3/6 fatty acids for reading in children: a randomized, double-blind, placebo-controlled trial in 9-year-old mainstream schoolchildren in Sweden. J Child Psychol Psychiatry. 2017 Jan;58(1):83-93. doi: 10.1111/jcpp.12614. Epub 2016 Aug 22. PMID 27545509